CLINICAL TRIAL: NCT05288127
Title: Phase II Study to Assess the Efficacy of Talazoparib in Asian Metastatic Breast Cancer Patients With a Homologous Recombinant Deficiency (HRD) Signature
Brief Title: Efficacy of Talazoparib in Asian Metastatic Breast Cancer Patients With a Homologous Recombinant Deficiency (HRD) Signature
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Collaborators: Cancer Research Malaysia (Other); Pfizer (Industry); Pantai Hospital Kuala Lumpur (Unknown); Hospital Sultan Ismail (Unknown)
Responsible Party: Principal Investigator, Ho Gwo Fuang, Professor Dr Ho Gwo Fuang, University of Malaya
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-CRM2020001
Record Dates: First submitted 2022-01-27; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: HRD 100 Gene Expression High; Triple Negative Breast Cancer
Keywords: Talazoparib; HRD 100 gene; Triple Negative Breast Cancer; BRCA 1/2
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Talazoparib Single Agent (Experimental): The study will have 1 treatment group. Patients will receive a single oral dose of talazoparib (Talzenna®) 1mg/day daily for 28-day cycles until progressive disease, limiting toxicities, intercurrent medical issues, patient withdrawal of consent, death, or end of trial whichever occurs first. Treatment will be administered on an outpatient basis. Talazoparib should be taken orally once daily (i.e., continuous daily dosing) at approximately the same time each day (preferably in the morning). Talazoparib will be swallowed whole and may be taken with or without food. If a subject vomits a dose, the subject should not take a second dose that calendar day. The subject should resume daily dosing the next day.
  Daily dosing of talazoparib can be interrupted for recovery from toxicity for up to 28 days. For interruptions longer than 28 days, treatment at the same or a reduced dose can be considered if the evidence of response or clinical benefit to talazoparib is noted.
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — The recommended dose is 1 mg talazoparib once daily. Patients should be treated until disease progression or unacceptable toxicity occurs. Daily dosing of talazoparib can be interrupted for recovery from toxicity for up to 28 days. For interruptions longer than 28 days, treatment at the same or a reduced dose can be considered based on the if evidence of response or clinical benefit to talazoparib is noted.
  Missing dose If the patient vomits or misses a dose, an additional dose should not be taken. The next prescribed dose should be taken at the usual time.
  Dose adjustments:
  To manage adverse drug reactions, interruption of treatment or dose reduction based on severity and clinical presentation should be considered.

SUMMARY:
This is an open label, non randomised, investigator-initiated Phase II study of single agent talazoparib (Talzenna®) in metastatic triple negative breast cancer patients with enriched HRD signature. Approximately 55 subjects will be enrolled in this study to examine the efficacy of talazoparib when given orally 1mg daily for days 1 to 28 for up to 28 months. The study will be conducted using the Simon two-stage phase II design, whereby this study will initially enroll 19 patients with RECIST v1.1 measurable disease with enriched HRD signature (stage I). There will be one interim analysis at the end of stage I and if 3 of the 19 have a response, then no further patient will be accrued. If 4 or more of the 19 patients have a response, then accrual would continue to stage II until a total of 55 patients have been enrolled. This study will be conducted in conformance with Good Clinical Practices. Specific procedures to be performed during the trial, as well as their prescribed times and associated visit windows, are outlined in the Trial Flow Chart.

DETAILED DESCRIPTION:
This is an open label, non randomised, investigator-initiated Phase II study of single agent talazoparib (Talzenna®) in metastatic triple negative breast cancer patients with enriched HRD signature. A total of 55 evaluable subjects will be enrolled in this study to examine the efficacy of talazoparib when given orally 1mg daily for days 1 to 28 for up to 28 months. The study will be conducted using the Simon two-stage phase II design, whereby this study will initially enroll 19 patients with RECIST v1.1 measurable disease with enriched HRD signature (stage I). There will be one interim analysis at the end of stage I and if 3 of the 19 have a response, then no further patient will be accrued. If 4 or more of the 19 patients have a response, then accrual would continue to stage II until a total of 55 patients have been enrolled. As it may take several weeks to determine if a patient has experienced a response, a temporary pause in the accrual to the trial may be necessary to ensure that enrollment to the second stage is warranted.

The purpose of this study is to determine if Talzenna® can help breast cancer patients who have not inherited an altered BRCA gene. We have identified a genetic signature called HRD100 which identifies patients who may respond to Talzenna®.

Disease status will be followed by imaging studies at interval of every 12 weeks, until disease progression, start of non-study treatment, withdrawal of consent to study participation, death or end of the study. RECIST 1.1 will be used as the primary endpoint of the response rate. Safety will be monitored according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Appendix 2).

Study Treatment will continue until any of the following occurs:

1. Disease progression, as defined by Response Evaluation Criteria in Solid Tumour (RECIST version 1.1);
2. Unacceptable toxicity;
3. Intercurrent illness that necessitates discontinuation of study treatment;
4. Investigator's decision to withdraw the subject,
5. Pregnancy;
6. Major violation to study treatment or procedure requirements;
7. Withdrawal of consent to treatment;
8. Death;
9. End of the study;
10. Other administrative reasons requiring cessation of study treatment.

Specific procedures to be performed during the trial, as well as their prescribed times and associated visit windows, are outlined in the SCHEDULE OF ACTIVITIES (SoA).

The study will be conducted in conformance with Good Clinical Practices.

The primary objective of the trial is to determine the objective response rate (CR+PR) of the single agent talazoparib in metastatic TNBC patients with enriched HRD signature using RECIST 1.1. Secondary Objective is to determine the progression free survival (PFS) and overall survival (OS) of talazoparib in metastatic TNBC patients.

Exploratory Objectives is to evaluate the HRD signature(s) in predicting response to PARP inhibitor in metastatic TNBC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures (including if needed to undergo germline BRCA testing and counselling as per local hospital practice) and availability for the duration of the study.
3. Women, aged 18 and above.
4. Received either one or two prior systemic treatments for metastatic breast cancer.
5. Histologically confirmed metastatic or recurrent triple-negative breast cancer (defined as ER <1%, PR <1%, HER2 negative, as per ASCO CAP guidelines).
6. Documented disease progression on the most recent therapy.
7. Have availability of 10 ml blood for germline BRCA testing if previous record of germline BRCA mutation status is not available.
8. If germline BRCA 1 or 2 (1/2) mutation positive, should be among the 5 patients (in Stage I) or 9 patients (in Stage II) with germline BRCA 1/2 mutation positive.
9. Can provide archival tumor tissue sample. Note: Formalin-fixed, paraffin embedded (FFPE) tissue blocks or tissues sections (>30% neoplastic cells, 2 x 10µm tissue curls each in 2 sterile 1.5ml-micro-centrifuge tubes) and 10 unstained slides are needed.
10. Can provide one 10ml and one 6-ml blood samples for future biomedical research.
11. Has classification as HRD High based on the HRD 100 gene expression analysis (Appendix 4)
12. Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Appendix 1).
13. Has adequate organ function as defined below: • Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ×upper limit of normal (ULN); if liver function abnormalities are due to hepatic metastasis, then AST and ALT ≤ 5 × ULN

    * Total serum bilirubin ≤ 1.5 × ULN (≤ 3 × ULN for Gilbert's syndrome)
    * Calculated creatinine clearance ≥ 30 mL/min by local laboratory or Cockcroft-Gault formula
    * Hemoglobin ≥ 9.0 g/dL with last transfusion at least 14 days before randomization
    * Absolute neutrophil count (ANC) ≥ 1500/mm3
    * Platelet count ≥ 100,000/mm3
14. Females of childbearing potential must be willing to use adequate contraception for the course of the study through at least 7 months after the last dose of study drug.
15. Patient must be able to swallow pills.

Exclusion Criteria:

1. Has ER-positive or PR-positive breast cancer.
2. Has HER2-positive breast cancer.
3. Have received prior treatment with a PARP inhibitor
4. Is currently on strong P-glycoprotein inhibitors.
5. Is germline BRCA 1/2 mutation carrier after the quota of germline BRCA 1/2 mutation carrier (inclusion criteria 4.1.7) of this trial have been fulfilled.
6. Has other malignancy that is either active or for which patients have received treatment within the last 5 years excluding non-melanoma skin cancer and carcinoma in situ of cervix
7. Have received platinum may not have relapsed within 6 months of the last dose of prior platinum therapy. For patients who have received platinum, at least 6 months must have elapsed between the last dose of platinum-based treatment and enrollment.
8. Is currently participating and receiving study therapy, or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study drug.
9. Has a known history of Human Immunodeficiency Virus (HIV).
10. Has known active Hepatitis B or Hepatitis C.
11. Has an active infection requiring systemic therapy.
12. Has significant cardiovascular disease, such as: History of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months;
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
14. Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit through at least 7 months after the last dose of study drug.
15. Has a known hypersensitivity to the components of the study drug or its analogs.
16. Known active brain metastases and/or carcinomatous meningitis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on gender identity.
Enrollment: 55 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Overall Responsive Rate (ORR) as assessed in RECIST 1.1 | [Time Frame: up to 28 months]
  It is commonly used in clinical trials to evaluate cancer treatments for objective response in solid tumors. The observed effect is attributable directly to the drug, not the natural history of the disease. Its application in tumor progression measurement is well accepted by regulatory authorities.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) using Kaplan-Meier (KM) method | [Time Frame: up to 28 months]
  PFS measure the time front start of study medication until the first sign of disease progression based on RECIST 1.1 or death from any cause, whichever occurs first. It is widely accepted endpoint in breast cancer Phase II clinical trials.
Overall Survival (OS) using Kaplan-Meier (KM) method | [Time Frame: up to 28 months]
  OS measures the date from study commencement to the date death from any cause. Patients alive or lost to follow up are censored. Overall survival as an endpoint is easily measured, unambiguous, objective and unaffected by the timing of assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Gwo Fuang Ho, FRCR, Principal Investigator — University of Malaya
Locations (1):
- University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia